CLINICAL TRIAL: NCT03997552
Title: Non-Incised Papillae Surgical Approach (NIPSA) Versus Marginal Approach by Palatal Incision and Minimally Invasive Surgical Technique (MIST) in Periodontal Regeneration: a Ramdomized Clinical Trial
Brief Title: NIPSA Versus Marginal Approach by Palatal Incision and MIST in Periodontal Regeneration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Antonio José Ortiz Ruiz, MD, Professor and researcher, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2409/2019
Record Dates: First submitted 2019-06-21; First posted 2019-06-25 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Periodontitis; Periodontal Diseases; Periodontal Pocket
MeSH Terms: conditions — Periodontitis; Periodontal Diseases; Periodontal Pocket

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-incised papillae surgical approach (NIPSA) (Experimental): To access the defect, a single horizontal or oblique apical incision will be made in the mucosa located on the bony cortex, far from the marginal tissues and apically to the edge of the bony crest delimiting the defect. The incision will be extended mesiodistally as necessary to allow access to the defect and correct debridement of the granulation tissue. The tissue coronal to the incision will be raised full thickness, trying to maintain the preoperative papillae architecture intact. The granulation tissue and epithelium of the pocket will be eliminated. The affected root will be scaled and planed, and calculus eliminated. Once the defect will be debrided, the enamel matrix derivates will be applied. Then the incision line will be sutured by a double suture line to facilitate closing without tension: The first with internal horizontal mattress sutures to approximate the connective tissue of both edges of the mucosal incision, and the second with single interrupted sutures.
  Interventions: Procedure: Non-incised papillae surgical approach (NIPSA)
- marginal approach by palatal incision (Active Comparator): A small incision in the palatal aspect and a limited papila elevation to the buccal aspect will be made for treating isolated periodontal defect. Enamel matrix derivates will be applied on the debrided root surfaces.
  Interventions: Procedure: marginal approach by palatal incision
- Minimally invasive surgical technique (MIST) (Active Comparator): The incision of the defect-associated papilla will be performed according to the principles of the papilla preservation techniques. Enamel matrix derivates will be applied on the debrided root surfaces. Stable primary closure of the flaps will be obtained with internal modified mattress sutures.
  Interventions: Procedure: Minimally invasive surgical technique (MIST)

INTERVENTIONS:
Procedure: Non-incised papillae surgical approach (NIPSA) — Periodontal reconstructive surgery
  Arms: Non-incised papillae surgical approach (NIPSA)
Procedure: marginal approach by palatal incision — Periodontal reconstructive surgery
  Arms: marginal approach by palatal incision
Procedure: Minimally invasive surgical technique (MIST) — Periodontal reconstructive surgery
  Arms: Minimally invasive surgical technique (MIST)

SUMMARY:
Three techniques for periodontal reconstruction will be compared, in which marginal access versus apical access will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with periodontitis.
* plaque index and bleeding index of < 30%.
* periodontal lesions with pocket probing depth > 5 mm.
* intrabony defect > 3 mm.
* intrabony defect configuration including a 1 and/or 2-wall component, always involving the buccal wall.

Exclusion Criteria:

* patients with systemic diseases that contraindicated treatment.
* third molars.
* teeth with incorrect endodontic or restorative treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-09-06 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Probing pocket depth (PD) | 12 months
  Probing pocket depth will be assessed with a periodontal probe, measured in mm from the gingival margin to the bottom of the pocket
Clinical attachment level (CAL) | 12 months
  Clinical attachment level will be assessed with a periodontal probe, measured in mm from the cementoenamel junction (CEJ) to the bottom of the pocket.
Recession (REC) | 12 months
  Recession, will be assessed with a periodontal probe, measured in mmm on the buccal aspect, from the CEJ to the gingival margin zenith.
Location of the tip of the papillae (TP) | 12 months
  Location of the tip of the papillae. Taking as reference the level of the mid-axis of the tooth, will be measured the distance from the CEJ at the zenith of the tooth to the tip of the papilla. A positive value will be recorded when the tip of the papillae is located coronally to the CEJ and a negative value otherwise.
  This outcome will be assessed with a periodontal probe and measured in mmm.
Keratinized tissue width (KT) | 12 months
  Keratinized tissue width will be assessed with a periodontal probe, measured in mm on the buccal aspect, from the gingival margin to the mucogingival line.
Bleeding on probing | 12 months
  Bleeding on probing could be positive or negative.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Odontologico Del Sureste Slp, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moreno Rodriguez JA, Ortiz Ruiz AJ, Caffesse RG. Periodontal reconstructive surgery of deep intraosseous defects using an apical approach. Non-incised papillae surgical approach (NIPSA): A retrospective cohort study. J Periodontol. 2019 May;90(5):454-464. doi: 10.1002/JPER.18-0405. Epub 2018 Nov 28. PMID 30421495
- [Result] Moreno Rodriguez JA, Ortiz Ruiz AJ, Caffesse RG. Supra-alveolar attachment gain in the treatment of combined intra-suprabony periodontal defects by non-incised papillae surgical approach. J Clin Periodontol. 2019 Sep;46(9):927-936. doi: 10.1111/jcpe.13158. Epub 2019 Jul 22. PMID 31190409